CLINICAL TRIAL: NCT01414569
Title: High Dose Dexamethasone as Pain Treatment After Arthroscopic Shoulder Surgery: A Randomised, Blinded Clinical Trial
Brief Title: Dexamethasone for Pain After Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Central Denmark Region (Other); The Hede Nielsen Family Foundation (Other); The Danish Rheumatism Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KTB-002; 2011-003082-15 (EudraCT Number)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Shoulder Impingement Syndrome; Arthritis
MeSH Terms: conditions — Shoulder Impingement Syndrome; Arthritis | interventions — Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 8 mg dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo, saline (Placebo Comparator)
  Interventions: Drug: Dexamethasone
- 40 mg dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Singe dose preoperatively in 100 ml saline intravenously
  Other Names: Fortecortin

SUMMARY:
The purpose of this study is to determine if a dose of 40 mg dexamethasone is more effective as pain treatment than the currently used dose of 8 mg after arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic subacromial decompression and/or acromioclavicular resection
* General anaesthesia
* Daysurgery, Horsens Hospital

Exclusion Criteria:

* Incompetent
* Pregnant
* Age under 18 or over 90 years
* Allergy toward dexamethasone
* Diabetes
* Active gastric ulcer
* Untreated hypertension
* Glaucoma
* Daily use of glucocorticoids or strong opioids
* Daily use of analgesics for unrelated illness
* Myasthenia gravis
* Mitochondrial disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain score by numeric rating scale | At 8 hours postoperatively

SECONDARY OUTCOMES:
Use of analgesics | During hospital stay, about 4 hours
  Need for supplemental analgesic medication during stay in recovery on the day of operation, until discharge.
Pain score by numeric rating scale | At about 8 a.m. on the first postoperative day
  On the morning of the first postoperative day, the self-evaluated level of pain as assessed by numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Bjørnholdt, MD, Principal Investigator — Aarhus University, Horsens Hospital; Kjeld Søballe, Prof. dr.med., Study Chair — Aarhus University Hospital; Lone Nikolajsen, ph.d., MD, Study Chair — Aarhus University Hospital
Locations (1):
- Horsens Hospital, Horsens, Denmark

REFERENCES:
- [Derived] Bjornholdt KT, Monsted PN, Soballe K, Nikolajsen L. Dexamethasone for pain after outpatient shoulder surgery: a randomised, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2014 Jul;58(6):751-8. doi: 10.1111/aas.12333. Epub 2014 May 13. PMID 24825530